CLINICAL TRIAL: NCT07019428
Title: Clinical Evaluation of a Modified Technique for Free Gingival Graft Stabilization Using Titanium Fixation Tacs Around Implants Versus Conventional Suturing Technique: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of a Modified Technique for Free Gingival Graft Stabilization Using Titanium Fixation Tacs Around Implants Versus Conventional Suturing Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Atef Kamal Ibrahim, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TacFGG
Record Dates: First submitted 2025-01-02; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Free Gingival Graft; Soft Tissue Augmentation Around Dental Implants; Inadequate Keratinized Tissue Around Dental Implants
Keywords: Free gingival graft; Titanium tacks; Keratinized tissue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free gingival graft stabilized by sutures (Active Comparator)
  Interventions: Procedure: Free gingival graft stabilized by sutures
- Free gingival graft stabilized by by Titanium fixation tacs (Experimental)
  Interventions: Procedure: Free gingival graft stabilized by Titanium fixation tacs

INTERVENTIONS:
Procedure: Free gingival graft stabilized by Titanium fixation tacs — Free gingival graft stabilized by Titanium fixation tacs , in patients with inadequate keratinized gingiva
  Arms: Free gingival graft stabilized by by Titanium fixation tacs
Procedure: Free gingival graft stabilized by sutures — Free gingival graft stabilized by sutures , in patients with inadequate keratinized gingiva
  Arms: Free gingival graft stabilized by sutures

SUMMARY:
The aim of this randomized, controlled, parallel-grouped, clinical trial is to evaluate the width of keratinized gingiva after free gingival graft stabilized by titanium fixation tacs compared to traditional suturing.

Research question:

In patients with inadequate keratinized gingiva undergoing soft tissue augmentation by free gingival graft , will graft stabilization using Titanium fixation tacs affect the amount of keratinized tissue gain compared to graft stabilization using sutures ?

DETAILED DESCRIPTION:
Free gingival graft obtained from the palate, usually replaces missing or lost keratinized tissue. Although it represents the gold standard, its success relies on providing intimate and atraumatic stabilization, as maintaining the plasmatic circulation is crucial for graft healing and perfusion, considering that judging the success of free gingival graftis based on the extent of the postoperative healing contraction and the quality of graft adherence to the underlying periosteum.

Suturing can be time consuming and sometimes fail to achieve a positive result. Also it was reported that for every one-minute increase of the gingival augmentation procedure time, there is a 4% likely increase for pain and a 3% for swelling.

However, by using fixation tacs the surgical time can be significantly reduced and the procedure can be less technique sensitive.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals of age ≥ 18 to 40 years with absence of active periodontal disease.
* Having inadequate width of keratinized gingiva (< 2 mm).
* No systemic disease according to Modified Cornell Medical Index health questionnaire
* Non-smoker.
* Full mouth plaque index (PI) and full-mouth bleeding on probing (BOP) score of ≤ 15%.
* No malocclusion, crowding, fillings, missing or supernumerary mandibular anterior teeth.
* No blood-borne conditions.

Exclusion Criteria:

* Active orthodontic treatment.
* Previous periodontal surgery.
* Systemic disease.
* Use of blood thinners.
* Use of any drugs that might lead to gingival enlargement.
* Mucogingival stress, bruxism.
* Pregnancy or lactation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Width of keratinized gingiva | 6-month

SECONDARY OUTCOMES:
Surgery time | Perioperative
  time spent from the beginning to the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amr Zahran, Professor of Periodontology, Principal Investigator — Cairo University; Manar El Zanaty, lecturer of Periodontology, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

DOCUMENTS (3):
  • Study Protocol (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT07019428/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT07019428/SAP_001.pdf
  • Informed Consent Form (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT07019428/ICF_002.pdf